# **Cover Page**

Release Date: June 16, 2025

ClinicalTrials.gov ID: NCT07033585

Unique Protocol ID: ANDA219975 + ANDA220011

**Brief Title:** Generic Drugs (Dapagliflozin and Saxagliptin) Treat Type 2 Diabetes

Patients with Controlled Cancers (GD-T2D)

Official Title: Generic Drugs (Dapagliflozin and Saxagliptin) Treat Type 2 Diabetes

**Patients with Controlled Cancers** 

Secondary IDs: NPI-1831468511 [Registry ID: HHS, Health Care Provider Individual]

NPI-1023387701 [Registry ID: HHS, Health Care Provider Organization] FWA00015357 [Registry ID: HHS, Human Protections Administrator]

IORG0007849 [Registry ID: HHS, IORG] IRB00009424 [Registry ID: HHS, IRB] ANDA219975 [Registry ID: FDA, ANDA] ANDA220011 [Registry ID: FDA, ANDA] Our investigation (NCT07033585) will be conducted in compliance with the requirements for informed consent (21 CFR Part 50) as follows:

### 21CFR § 50.3 (f)

Sponsor-investigator means an individual who both initiates and actually conducts, alone or with others, a clinical investigation, i.e., under whose immediate direction the test article is administered or dispensed to, or used involving, a subject. The term does not include any person other than an individual, e.g., corporation or agency.

- 2020 Active Member, Fellow of the APCR (FAPCR), Academy of Physicians in Clinical Research (APCR) -APCR Membership Eligibility - Physician Investigator
  - Certificate of Fellow of Academy of Physicians in Clinical Research (FAPCR)
  - Academy of Physicians in Clinical Research (APCR)
    - ♦ PI (Principal Investigator) in clinical trials
    - **♦ Medical Director of Clinical Research Site**
- 2025-06 FDA Pre-Assignment IND 177776 for Type 2 Diabetes Oral Mix Prescription
  - Sponsor: HAN XU
- 2025-06 ClinicalTrials.gov ID: NCT07033585
  - Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair
  - Responsible Party: Sponsor-Investigator
  - Sponsor-Investigator: Han Xu, M.D., Ph.D., FAPCR
  - Study Principal Investigator [Principal Investigator (PI)]: Han Xu, M.D., Ph.D., FAPCR

In FDA IND Pre-Assignment, I (HAN XU) am Sponsor. In my APCR documents, Han Xu, M.D., Ph.D., FAPCR had been defined as PI (Principal Investigator) in clinical trials. In my document ClinicalTrials.gov ID: NCT07033585, I (Han Xu, M.D., Ph.D., FAPCR) am defined as Responsible Party (Sponsor-Investigator). So, I must be the sponsor-investigator (S-I) of my clinical trial. And I (Han Xu, M.D., Ph.D. i.e., Sponsor i.e., Sponsor-Investigator) can both initiate and conduct, alone or with others, my clinical investigation. At the same time, I am a qualified investigator for my ANDA type 2 diabetes clinical trial.

### 21 CFR § 50.20 -- General requirements for informed consent.

Except as provided in §50.23 and §50.24, no investigator may involve a human being as a subject in research covered by these regulations unless the investigator has obtained the legally effective informed consent of the subject or the subject's legally authorized representative. An investigator shall seek such consent only under circumstances that provide the prospective subject or the representative sufficient opportunity to consider whether or not to participate and that minimize the possibility of coercion or undue influence. The information that is given to the subject or the representative shall be in language understandable to the subject or the representative. No informed consent, whether oral or written, may include any exculpatory language through which the subject or the representative is made to waive or appear to waive any of the subject's legal rights, or releases or appears to release the investigator, the sponsor, the institution, or its agents from liability for negligence.

### 21 CFR § 50.25 -- Elements of informed consent.

- (a) Basic elements of informed consent. In seeking informed consent, the following information shall be provided to each subject:
- (1) A statement that the study involves research, an explanation of the purposes of the research and the expected duration of the subject's participation, a description of the procedures to be followed, and identification of any procedures which are experimental.
  - (2) A description of any reasonably foreseeable risks or discomforts to the subject.
- (3) A description of any benefits to the subject or to others which may reasonably be expected from the research.
- (4) A disclosure of appropriate alternative procedures or courses of therapy, if any, that might be advantageous to the subject.

- (5) A statement describing the extent, if any, to which confidentiality of records identifying the subject will be maintained and that notes the possibility that the Food and Drug Administration may inspect the records.
- (6) For research involving more than minimal risk, an explanation as to whether any compensation and an explanation as to whether any medical therapys are available if injury occurs and, if so, what they consist of, or where further information may be obtained.
- (7) An explanation of whom to contact for answers to pertinent questions about the research and research subjects' rights, and whom to contact in the event of a research-related injury to the subject.
- (8) A statement that participation is voluntary, that refusal to participate will involve no penalty or loss of benefits to which the subject is otherwise entitled, and that the subject may discontinue participation at any time without penalty or loss of benefits to which the subject is otherwise entitled.
- (b) Additional elements of informed consent. When appropriate, one or more of the following elements of information shall also be provided to each subject:
- (1) A statement that the particular therapy or procedure may involve risks to the subject (or to the embryo or fetus, if the subject is or may become pregnant) which are currently unforeseeable.
- (2) Anticipated circumstances under which the subject's participation may be terminated by the investigator without regard to the subject's consent.
  - (3) Any additional costs to the subject that may result from participation in the research.
- (4) The consequences of a subject's decision to withdraw from the research and procedures for orderly termination of participation by the subject.
- (5) A statement that significant new findings developed during the course of the research which may relate to the subject's willingness to continue participation will be provided to the subject.
  - (6) The approximate number of subjects involved in the study.
- (c) When seeking informed consent for applicable clinical trials, as defined in 42 U.S.C. 282(j)(1)(A), the following statement shall be provided to each clinical trial subject in informed consent documents and processes. This will notify the clinical trial subject that clinical trial information has been or will be submitted for inclusion in the clinical trial registry databank under paragraph (j) of section 402 of the Public Health Service Act. The statement is: "A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time."
- (d) The informed consent requirements in these regulations are not intended to preempt any applicable Federal. State, or local laws which require additional information to be disclosed for informed consent to be legally effective.
- (e) Nothing in these regulations is intended to limit the authority of a physician to provide emergency medical care to the extent the physician is permitted to do so under applicable Federal, State, or local law.

## 21 CFR § 50.27 Documentation of informed consent.

- (a) Except as provided in §56.109(c), informed consent shall be documented by the use of a written consent form approved by the IRB and signed and dated by the subject or the subject's legally authorized representative at the time of consent. A copy shall be given to the person signing the form.
  - (b) Except as provided in §56.109(c), the consent form may be either of the following:
- (1) A written consent document that embodies the elements of informed consent required by §50.25. This form may be read to the subject or the subject's legally authorized representative, but, in any event, the investigator shall give either the subject or the representative adequate opportunity to read it before it is signed.

(2) A short form written consent document stating that the elements of informed consent required by §50.25 have been presented orally to the subject or the subject's legally authorized representative. When this method is used, there shall be a witness to the oral presentation. Also, the IRB shall approve a written summary of what is to be said to the subject or the representative. Only the short form itself is to be signed by the subject or the representative. However, the witness shall sign both the short form and a copy of the summary, and the person actually obtaining the consent shall sign a copy of the summary. A copy of the summary shall be given to the subject or the representative in addition to a copy of the short form.

# **Contents**

| Phase 2 ANDA Type 2 Diabetes Study Consent Form | 4 |
|---|---|
| Study Title for Study Participants: | ∠ |
| Official Study Title for Internet Search on http://www.ClinicalTrials.gov: | ∠ |
| What is the usual approach to your type 2 diabetes? | |
| What are my other choices if I do not take part in this study? | ∠ |
| Why is this study being done? | 5 |
| What are the study groups? | |
| How long will I be in this study? | 5 |
| What extra tests will I have if I take part in this study? | <i>6</i> |
| What possible risks can I expect from taking part in this study? | <i>6</i> |
| What possible benefits can I expect from taking part in this study? | |
| Can I stop taking part in this study? | |
| What are my rights in this study? | |
| What are the costs of taking part in this study? | |
| What happens if I am injured or hurt because I took part in this study? | |
| Who will see my medical information? | 8 |
| Where can I get more information? | 8 |
| Who can answer my questions about this study? | 8 |
| ADDITIONAL STUDIES SECTION: | 8 |
| This section is about an optional study you can choose to take part in | 8 |
| My Signature Agreeing to Take Part in the Main Study | 11 |

#### 21 CFR 312.23(a)(1)(v)

A commitment to conduct the investigation in accordance with all other applicable regulatory requirements.

#### 21 CFR 312.53(c)(1)(vi)(d)

Will inform any potential subjects that the drugs are being used for investigational purposes and will ensure that the requirements relating to obtaining informed consent (21 CFR part 50) and institutional review board review and approval (21 CFR part 56) are met:

#### Statement

I write the <u>commitment</u> with respect to each clinical study involving human subjects that it either will be conducted in compliance with the institutional review board regulations in part 56 or will not be subject to the regulations under §56.104 or §56.105; and that it either will be conducted in compliance with the informed consent regulations in part 50 or will not be subject to the regulations under §50.23 and §50.24.

Generic Drugs Treat Type 2 Diabetes Patients with Controlled Cancers

- Usual Approach Group -- Generic Drugs Oral Mix Prescription 1
- Study Approach Group -- Generic Drugs Oral Mix Prescription 2

The investigation (NCT07033585) will be conducted in compliance with the requirements for 21 CFR Part 56 as follows:

### 21 CFR § 56.102 (k)

Sponsor-investigator means an individual who both initiates and actually conducts, alone or with others, a clinical investigation, i.e., under whose immediate direction the test article is administered or dispensed to, or used involving, a subject. The term does not include any person other than an individual, e.g., it does not include a corporation or agency. The obligations of a sponsor-investigator under this part include both those of a sponsor and those of an investigator.

I (sponsor-investigator) will actually conduct, with online referral clinical investigators, the clinical investigation (NCT07033585), i.e., under whose immediate direction the test article is administered or dispensed to, or used involving, a subject.

Our investigation (NCT07033585) will be conducted in compliance with the requirements for **21 CFR Part 50** as follows:

#### 21 CFR § 50.3 (f)

Sponsor-investigator means an individual who both initiates and actually conducts, alone or with others, a clinical investigation, i.e., under whose immediate direction the test article is administered or dispensed to, or used involving, a subject. The term does not include any person other than an individual, e.g., corporation or agency.

I (sponsor-investigator) will actually conduct, with online referral clinical investigators, the clinical investigation (NCT07033585), i.e., under whose immediate direction the test article is administered or dispensed to, or used involving, a subject.

## Phase 2 ANDA Type 2 Diabetes Study Consent Form

## **Study Title for Study Participants:**

Generic Drugs Treat Type 2 Diabetes Patients with Controlled Cancers (GD-T2D)

## Official Study Title for Internet Search on http://www.ClinicalTrials.gov:

Study 00001 - (NCT07033585) - ANDA Clinical Study -- Generic Drugs Treat Type 2 Diabetes Patients with Controlled Cancers.

**LABEL:** FARXIGA - dapagliflozin tablet, film coated (<a href="https://dailymed.nlm.nih.gov">https://dailymed.nlm.nih.gov</a>) **LABEL:** ONGLYZA - saxagliptin tablet, film coated (<a href="https://dailymed.nlm.nih.gov">https://dailymed.nlm.nih.gov</a>)

LABEL: METFORMIN HYDROCHLORIDE - metformin tablet (https://dailymed.nlm.nih.gov)

Nan Fang Yi Ke Da Xue Xue Bao: 2019 Nov 30; 39(11): 1305-1311.

## What is the usual approach to your type 2 diabetes?

You are being asked to take part in this research study because you have had diagnosis for your type 2 diabetes. People who are not in a research study may be treated with generic drugs after diagnosis. There are FDA-approved drugs (Dapagliflozin plus Saxagliptin plus Metformin Oral Mix Prescription) (Mix-1) (Mix-2) that are commonly used. For patients who receive the usual approach for this diabetes about 70 out of 100 may be controlled of diabetes in one year.

# What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. For example:

- you may choose to have the usual approach described above ...
- you may choose to take part in a different study if one is available ...
- or you could decide not to be treated for diabetes ...

# Why is this study being done?

The purpose of this study is to test any good and bad effects of the study therapy dose Oral Mix Prescription - 2 compared to the usual therapy dose Oral Mix Prescription - 1. The study group drugs could cause therapeutic effects of therapy by preventing your diabetes from returning or they could cause side effects or reduce the benefits of therapy. This study will allow the researchers to know whether the study therapy drugs are better, the same or worse than not doing so. Record using generic drugs therapeutic effects and side effects of treating type 2 diabetes, based on laboratory test. The therapy efficacy can arrive at a higher level. The therapy risk can arrive at a lower level. There will be about 600 people taking part in this study.

## What are the study groups?

This study has two study groups.

- Group 1 will get the usual dose generic drugs to treat type 2 diabetes:
  - Oral Mix Prescription 1 (12 weeks):
  - ✓ NDC 0310-6210-30 (FARXIGA dapagliflozin tablet, film coated) -- 10 mg orally once daily
  - ✓ NDC 0310-6105-30 (ONGLYZA saxagliptin tablet, film coated) -- 5 mg orally once daily
  - ✓ NDC 65162-175-10 (METFORMIN HYDROCHLORIDE metformin tablet) -- 500 mg twice a day
  - o This therapy will be for 90 days.
- Group 2 will get the study dose generic drugs to treat type 2 diabetes:
  - Oral Mix Prescription 2 (12 weeks):
  - ✓ China Import dapagliflozin tablet (ANDA 219975) -- 10 mg orally once daily
  - ✓ China Import saxagliptin tablet (ANDA 220011) -- 5 mg orally once daily
  - ✓ NDC 65162-175-10 (METFORMIN HYDROCHLORIDE metformin tablet) -- 500 mg twice a day
  - o This therapy will be for 90 days.

A computer will by chance assign you to therapy groups in the study. This is called randomization. This is done by chance because no one knows if one study group is better or worse than the other. Neither you nor your doctor can choose which group you will be in.

Another way to find out what will happen to you during this study is to read the chart below. Start reading on the left side and read across to the right, following the lines and arrows.



# How long will I be in this study?

You will receive the study drugs for six months if you are in Group 1 and in Group 2. After you finish the study drugs, you will be asked to see your study doctor for follow-up examinations for 2 years. Your study doctor would like to continue to watch you for side effects and follow your condition for the rest of your life.

# What extra tests will I have if I take part in this study?

If you are assigned to Group 1, all of the tests you will have been part of the usual approach to your diabetes. If you are assigned to Group 2, all of the tests you will have been part of the study approach for your diabetes. There are blood, urine, and gene tests that you will need to have:

- Detect Hemoglobin A1c (HbA1c)
- Detect fasting blood glucose (FBG)
- Detect 2-hour postprandial blood glucose (2 hPBG)
- Detect fasting insulin (FINS)
- Detect 2-hour postprandial insulin (2 hPINS)
- If you have an allergic reaction to type 2 diabetes drugs, you will have an extra blood test.
- You will need urine tests every week while you are taking type 2 diabetes drugs.
- You will need blood tests every week while you are taking type 2 diabetes drugs.

Your insurance company will be charged for the blood, urine, biopsy, and gene tests related to oncology drugs.

# What possible risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work or home and spend more time in the hospital or doctor's office than usual.
- You may be asked sensitive or private questions which you normally do not discuss.
- The generics drugs may not be better, and could be possibly worse, than receiving the other drugs.

The study drugs used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood, urine, and genes, and will let you know if changes occur that may affect your health. There is also a risk that you could have side effects from the usual chemotherapy drugs and the study chemotherapy drugs.

Here are important points about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.

Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different so they can see if you have a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.

The tables below show the most common and the most serious side effects that researchers know about. There might be other side effects that researchers do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

Study Group 1 and Group 2 - Possible Side Effects of the usual therapy and the study therapy for this type 2 diabetes:

- LABEL: FARXIGA dapagliflozin tablet, film coated (NDA202293) (https://dailymed.nlm.nih.gov)
- LABEL: ONGLYZA saxagliptin tablet, film coated (NDA022350) (https://dailymed.nlm.nih.gov)
- LABEL: METFORMIN HYDROCHLORIDE metformin tablet (ANDA077880) (https://dailymed.nlm.nih.gov)

Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

Reproductive risks: You should not get pregnant, breastfeed, or father a baby while in this study. The drugs used in this study could be very damaging to an unborn baby. Check with the study doctor about what types of birth control, or pregnancy prevention, to use while in this study.

# What possible benefits can I expect from taking part in this study?

It is not possible to know at this time if the study therapy is better than the usual therapy, so this study may or may not help you. This study will help researchers learn things that will help people in the future.

# Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information to the organization running the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If new information becomes available
- If you do not follow the study rules
- If the study is stopped by the sponsor, IRB, or FDA

# What are my rights in this study?

Taking part in this study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care or any legal rights.

For questions about your rights while in this study, call the <u>Medicine Invention Design, Inc.</u> Institutional Review Board (IRB) at <u>1-301-222-7143.</u>

# What are the costs of taking part in this study?

The usual therapy drugs and the study therapy drugs will be supplied at charge by your insurance company while you take part in this study. The cost of getting the drugs ready and giving them to you is not provided by you so your insurance company will have to pay for this. It is possible that the usual therapy drugs and the study therapy drugs may not continue to be supplied while you are on the study. Although not likely, if this occurs, your study doctor will talk to you about your options.

Your health plan / insurance company will need to pay for all of the other costs of treating your diabetes while in this study, including the cost of managing any side effects. Before you decide to be in the study, you should check with your health plan or insurance company to find out exactly what they will pay for.

You will not be paid for taking part in this study.

# What happens if I am injured or hurt because I took part in this study?

If you are injured or hurt as a result of taking part in this study and need medical therapy, please tell your study doctor. The study sponsors will not offer to pay for medical therapy for injury. Your insurance company may be willing to pay for study-related injury. If you have no insurance, you will be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive some help with this even though you participate in the study.

# Who will see my medical information?

Your privacy is very important to us, and the researchers will make every effort to protect it. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you. Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- The Medicine Invention Design, Inc. and other drug companies support this study.
- The Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting the people who take part in the study.
- The Food and Drug Administration in the U.S. and similar agencies in other countries involved in the study.

# Where can I get more information?

You may visit the Web page at <a href="https://clinicaltrials.gov/ct2/show/NCT07033585">https://clinicaltrials.gov/ct2/show/NCT07033585</a> for more information about this study. You may also call the Diabetes Information Service of the Medicine Invention Design, Inc. to get the same information at: 1-301-222-7143.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## Who can answer my questions about this study?

You can talk to the study doctor about any questions or concerns you have about this study or to report side effects or injuries. Contact the study doctors via <a href="Han Xu, M.D.">Han Xu, M.D.</a>, <a href="Ph.D.">Ph.D.</a>, <a href="IRB Chair">IRB Chair</a>, <a href="Sponsor-Investigator">Sponsor-Investigator</a>, <a href="IORG Director">IORG Director</a> at <a href="1-301-222-7143">1-301-222-7143</a>.

## **ADDITIONAL STUDIES SECTION:**

# This section is about an optional study you can choose to take part in

You can still take part in the main study even if you say 'no' to this study. If you sign up for but cannot complete this study for any reason, you can still take part in the main study.

## **Optional Sample Collections for Biobanking for Possible Future Studies**

Researchers are trying to learn more about cancer, diabetes, and other health problems. Much of this research is done using samples from your genes, blood, urine, or other fluids. Through these studies, researchers hope to find new ways to prevent, detect, treat, or cure health problems.

Some of these studies may be about genes. Genes carry information about features that are found in you and in people who are related to you. Researchers are interested in the way that genes affect how your body responds to therapy.

The researchers ask your permission to store and use your samples and health information for medical research. The research that may be done is unknown at this time. Storing samples for future studies is called 'biobanking'. The Biobank is being run by the MIDINC Clinical Research Multiple Group and supported by the Medicine Invention Design, Inc. (MIDI).

#### What is involved?

If you agree to take part, here is what will happen next:

- 1) A sample from the gene that was collected at the time of your blood will be sent to the Biobank.
- 2) Your sample and some related information may be stored in the Biobank along with samples and information from other people who take part. The samples will be kept until they are used up.
- 3) Qualified researchers can submit a request to use the materials stored in the Biobank. A science committee at the clinical trials organization, and/or the MIDI, will review each request. There will also be an ethics review to ensure that the request is necessary and proper. Researchers will not be given your name or any other information that could directly identify you.
- 4) Neither you nor your study doctor will be notified when research will be conducted or given reports or other information about any research that is done using your samples.
- 5) Some of your genetic and health information may be placed in central databases that may be public, along with information from many other people. Information that could directly identify you will not be included.

## What are the possible risks?

- 1) There is a risk that someone could get access to the personal information in your medical records or other information the researchers have stored about you.
- 2) There is a risk that someone could trace the information in a central database back to you. Even without your name or other identifiers, your genetic information is unique to you. The researchers believe the chance that someone will identify with you is very small, but the risk may change in the future as people come up with new ways of tracing information.
- 3) In some cases, this information could be used to make it harder for you to get or keep a job or insurance. There are laws against the misuse of genetic information, but they may not give full protection. There can also be a risk in knowing genetic information. New health information about inherited traits that might affect you or your blood relatives could be found during a study. The researchers believe the chance these things will happen is very small but cannot promise that they will not occur.

### How will information about me be kept private?

Your privacy is very important to the researchers, and they will make every effort to protect it. Here are just a few of the steps they will take:

- 1) When your sample is sent to the researchers, no information identifying you (such as your name) will be sent. Samples will be identified by a unique code only.
- 2) The list that links the unique code to your name will be kept separate from your sample and health information. Any Biobank and MIDINC Clinical Research Multiple Group staff with access to the list must sign an agreement to keep your identity confidential.
- 3) Researchers to whom the MIDINC Clinical Research Multiple Group sends your sample, and information will not know who you are. They must also sign an agreement that they will not try to find out who you are.
- 4) Information that identifies you will not be given to anyone, unless required by law.
- 5) If research results are published, your name and other personal information will not be used.

## What are the possible benefits?

You will not benefit from taking part. The researchers, using the samples from you and others, might make discoveries that could help people in the future.

## Are there any costs or payments?

There are no costs to you or your insurance. You will not be paid for taking part. If any of the research leads to new tests, drugs, or other commercial products, you will not share in any profits.

## What if I change my mind?

If you decide you no longer want your samples to be used, you can call the study doctor on 1-301-222-7143 who will let the researchers know. Then, any sample that remains in the bank will no longer be used. Samples or related information that have already been given to or used by researchers will not be returned.

### What if I have more questions?

If you have questions about the use of your samples for research, contact the study doctor via 1-301-222-7143.

Please circle your answer to show whether or not you would like to take part in this optional biobanking study.

My samples and related information may be kept in a Biobank for use in future health research.

### YES NO

I agree that my study doctor, or their representative, may contact me or my physician to see if I wish to participate in other research in the future.

#### YES NO

This is the end of the section about optional studies.

### \*\*\*\*\*Note:

Based on FWA00015357, this Informed Consent Form (ICF) is written by Han Xu, M.D., Ph.D., Sponsor-Investigator. Also, this ICF is reviewed and approved by IRB00009424 and IORG0007849. If you need or find any changes to this ICF, please inform IRB, IORG, or Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, IRB Chair, IORG Director immediately.

**Phone:** +1-301-222-7143 **Fax:** +1-866-458-0099

**E-mail:** hanxumd@gmail.com

I write following <u>statement</u> with respect to each clinical study involving human subjects that it either will be conducted in compliance with the institutional review board regulations in **part 56** or will **not** be subject to the regulations under §56.104 or §56.105; and that it either will be conducted in compliance with the informed consent regulations in **part 50** or will **not** be subject to the regulations under §50.23 and §50.24.

Our investigation (NCT07033585) will be conducted in compliance with the requirements for 21 CFR Part 50 as follows:

### 21 CFR § 50.3 (f)

Sponsor-investigator means an individual who both initiates and actually conducts, alone or with others, a clinical investigation, i.e., under whose immediate direction the test article is administered or dispensed to, or used involving, a subject. The term does not include any person other than an individual, e.g., corporation or agency.

I (sponsor-investigator) will actually conduct, with online referral clinical investigators, the clinical investigation, i.e., under whose immediate direction the test article is administered or dispensed to, or used involving, a subject.

# My Signature Agreeing to Take Part in the Main Study

I have read this consent form, or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed copy of this form. I agree to take part in the main study and in the optional study if I have circled "Yes".

| Participant's signature |
|-------------------------------------|
| Date of signature |
| Study Doctor's signature |
| Date of signature |
| Study Nurse / Assistant's signature |
| Date of signature |